CLINICAL TRIAL: NCT02082067
Title: Total Knee Arthroplasty & Outcome: A Prospective Randomized Comparison Between Adductor Canal Block and Femoral Nerve Block
Brief Title: Total Knee Prosthesis With Continuous Block of Adductor Canal and Outcome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, Medical Doctor, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOGPGC05-14
Record Dates: First submitted 2014-02-28; First posted 2014-03-10 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Anesthesia, Spinal; Ketorolac; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adductor canal (Experimental): All patients in the arm will receive continuous adductor canal block under ultrasound guidance. 10ml of Ropivacaine 0,75%, BBraun, Germany, will be injected to dilate adductor canal. After catheter insertion 10ml of Ropivacaine 0,75% will be injected.
  Interventions: Procedure: Adductor canal; Procedure: Spinal Anesthesia; Procedure: Local anesthetic infusion; Procedure: Intravenous analgesia; Drug: Ropivacaine 0,75%; Drug: Levobupivacaine 0,5%; Drug: Levobupivacaine 0,125%; Drug: Ketorolac 30mg; Drug: Morphine; Device: stimulong sono, Pajunk, Germany
- Femoral (Active Comparator): All patients in the arm will receive continuous femoral nerve block under ultrasound guidance. Correct position of catheter will be check with injection of 20ml Ropivacaine 0,75% BBraun, Germany medial to femoral nerve.
  Interventions: Procedure: Femoral; Procedure: Spinal Anesthesia; Procedure: Local anesthetic infusion; Procedure: Intravenous analgesia; Drug: Ropivacaine 0,75%; Drug: Levobupivacaine 0,5%; Drug: Levobupivacaine 0,125%; Drug: Ketorolac 30mg; Drug: Morphine; Device: stimulong sono, Pajunk, Germany
- Controls (Placebo Comparator): No patients of this arm receive continuous nerve block. Intravenous opioids analgesia will be administered.
  Interventions: Procedure: Spinal Anesthesia; Procedure: Intravenous analgesia; Drug: Levobupivacaine 0,5%; Drug: Ketorolac 30mg; Drug: Morphine

INTERVENTIONS:
Procedure: Adductor canal — Perinervous catheter (stimulong sono- Pajunk, Germany) will be insert in adductor canal through tuohy needle (18G, 100mm length) under ultrasound guidance.
  Arms: Adductor canal
Procedure: Femoral — Perinervous catheter (stimulong sono- Pajunk, Germany) will be insert between femoral nerve and femoral artery through tuohy needle (18G, 100mm length) under ultrasound guidance.
  Arms: Femoral
Procedure: Spinal Anesthesia — Spinal anesthesia will be perform at L3-L4 or L4-L5 level. Levobupivacaine 0,5% 12mg will be injected.
Procedure: Local anesthetic infusion — Continuous infusion of levobupivacaine 0,125% at 8ml/h rate through perinervous catheter until 5th postoperative day.
  Arms: Adductor canal; Femoral
Procedure: Intravenous analgesia — Ketorolac 30mg 3 times/day and morphine Patients Control Analgesia (1mg/h, max 4mg/h) administered.
Drug: Ropivacaine 0,75%
  Arms: Adductor canal; Femoral
Drug: Levobupivacaine 0,5%
Drug: Levobupivacaine 0,125%
  Arms: Adductor canal; Femoral
Drug: Ketorolac 30mg
Drug: Morphine
Device: stimulong sono, Pajunk, Germany
  Arms: Adductor canal; Femoral

SUMMARY:
Aim of this study is to evaluate the effects of the adductor canal block on the early and medium term ( 1 month) rehabilitation compared to the continuous femoral block commonly used in the knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total knee arthroplasty

Exclusion Criteria:

* diabetes
* neurological disorders
* coagulation disorders
* rheumatoid arthritis
* chronic opioids therapy
* allergy to local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Up and Go test | 5th postoperative day
  Knee functional evaluation at 5th postoperative day. "up and go" test: time need to get up from a chair, walk for 3 meters, and come back to seat down on the chair

SECONDARY OUTCOMES:
VAS score | up to POD5
  Evaluation of VAS static and VAS dynamic during hospital stay
Morphine request | up to POD5
  Opioids consumption will be recorded throughout postoperative period
Range of motion | 5th postoperative day
  Physiotherapist measures the maximum active/passive range of motion
Falling risk | 5th postoperative day
  Evaluation of falling risk with Berg Balance Scale
Quadriceps strength | 5th postoperative day
  evaluate muscle strength with an isometric force dynamometer to measure the force produced during a maximum voluntary isometric contraction in a lying position by the knee flex to 90°.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Cappelleri, M.D., Principal Investigator — ASST Gaetano Pini-CTO
Locations (1):
- Istituto ortopedico Gaetano Pini, Milan, Italy